CLINICAL TRIAL: NCT01638923
Title: A Multicenter, Double-blind, Randomized, Parallel-group, Placebo-controlled, 7 Cycle Duration (196 Days), Phase 3 Study to Investigate the Efficacy and Safety of Oral Estradiol Valerate / Dienogest Tablets for the Treatment of Heavy Menstrual Bleeding
Brief Title: Study of a 4-phasic Oral Contraceptive for the Treatment of Heavy Menstrual Bleeding
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 91774; X311965 (Other: Company Internal)
Record Dates: First submitted 2012-06-20; First posted 2012-07-12 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Metrorrhagia
Keywords: Heavy Menstrual Bleeding; Efficacy; Safety; Oral contraceptive; Estradiol valerate; Dienogest
MeSH Terms: conditions — Metrorrhagia; Menorrhagia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: EV/DNG (Qlaira, Natazia, BAY86-5027)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: EV/DNG (Qlaira, Natazia, BAY86-5027) — 2 days of 3 mg estradiol valerate (EV);5 days of 2 mg EV + 2 mg dienogest (DNG);17 days of 2 mg EV + 3 mg DNG;2 days of 1 mg EV;2 days of placebo. A blister card consists of 28 pills, taken orally once a day for 7 cycles of 28 days each.
  Arms: Arm 1
Drug: placebo — Matching placebo to be taken orally daily for 7 cycles of 28 days each.
  Arms: Arm 2

SUMMARY:
To evaluate efficacy and safety of a combined oral contraceptive of estradiol valerate and dienogest in the treatment of heavy menstrual bleeding

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years or older in generally good health with a diagnosis of heavy menstrual bleeding without organic pathology, requesting contraception
* Willingness to use barrier contraception (e.g., condoms) from screening to study completion
* Willingness to use and collect sanitary protection (pads and tampons) provided by the sponsor and compatible with the alkaline hematin test throughout study completion

Exclusion Criteria:

* Current diagnosis of organic uterine bleeding
* History of endometrial ablation, or dilatation and curettage within 2 months of Visit 1.
* Clinically significant pelvic findings (whether or not confirmed by transvaginal ultrasound [TVU]).
* Clinically significant abnormal results of breast examination (breast palpation).
* Positive pregnancy test at Visit 1
* Less than three months since delivery, abortion, or lactation before to start Visit 1
* Other contraceptive methods
* Any disease or condition that may worsen under hormonal treatment
* Smokers over the age of 35
* Body mass index >32

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Absolute change in Menstrual Blood Loss (MBL) at baseline and 90 days | 90 day baseline period and 90 days during treatment period

SECONDARY OUTCOMES:
Proportion of subjects with successful treatment | 90 days during treatment phase
  Successful treatment is defined as no bleeding episode with MBL of 80 mL or more and a decrease to a value </=50% of MBL compared to 90 day run-in period
Percent change of MBL at baseline and 90 day period during treatment phase | Baseline and 90 days during treatment phase
Absolute change of average MBL at baseline and up to cycle 7 (one cycle = 28 days) | Baseline and cycle 1, cycle 2, cycle 3, cycle 4, cycle 5, cycle 6, cycle 7
Proportion of subjects with improvement in the investigator's global assessment scale on Day 84 | Treatment day 84
  Investigator's global assessment scale: 0 = not assessed; 1 = very much improved; 2 = much improved; 3 = improved; 4 = no change; 5 = worse; 6 = much worse; 7 = very much worse; Improvement is defined as the assessment score = 1, 2, or 3.
Proportion of subjects with improvement in the investigator's global assessment scale on Day 196 | Treatment day 196
  Investigator's global assessment scale: 0 = not assessed; 1 = very much improved; 2 = much improved; 3 = improved; 4 = no change; 5 = worse; 6 = much worse; 7 = very much worse; Improvement is defined as the assessment score = 1, 2, or 3.
Proportion of subjects with improvement in the subject's global assessment scale on Day 84 | Treatment day 84
  Subject's global assessment scale: 0 = not assessed; 1 = very much improved; 2 = much improved; 3 = improved; 4 = no change; 5 = worse; 6 = much worse; 7 = very much worse; Improvement is defined as the assessment score = 1, 2, or 3.
Proportion of subjects with improvement in the subject's global assessment scale on Day 196 | Treatment day 196
  Subject's global assessment scale: 0 = not assessed; 1 = very much improved; 2 = much improved; 3 = improved; 4 = no change; 5 = worse; 6 = much worse; 7 = very much worse; Improvement is defined as the assessment score = 1, 2, or 3.
Number of participants with adverse events as a measure of safety and tolerability | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (29):
- China (17):
  - Guangzhou, Guangdong
  - Nanning, Guangxi
  - Shijiazhuang, Hebei
  - Wuhan, Hubei
  - Changsha, Hunan
  - Hengyang, Hunan
  - Dalian, Liaoning
  - Shenyang, Liaoning
  - Xi'an, Shaanxi
  - Jinan, Shandong
  - Chengdu, Sichuan
  - Beijing
  - Changchun
  - Chongqing
  - Qingdao
  - Shanghai
  - Tianjin
- Philippines (2):
  - Manila
  - Quezon City
- Russia (5):
  - Irkutsk
  - Ivanovo
  - Krasnodar
  - Moscow
  - Saint Petersburg
- Singapore, Singapore
- Taiwan (3):
  - Taichung
  - Tainan
  - Taipei
- Bangkok, Thailand